CLINICAL TRIAL: NCT01821066
Title: A Phase 1 Open-Label Fixed-Sequence Two-Period Crossover Study Of The Effect Of Multiple Doses Of Tamoxifen On PD-0332991 Pharmacokinetics In Healthy Male Volunteers
Brief Title: A Study To Determine If Coadministration Of Tamoxifen Alters The Extent Or Rate Of Palbociclib (PD-0332991) Absorption Or Elimination In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A5481026
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: PD-0332991; palbociclib; tamoxifen; drug-drug interaction (DDI) study
MeSH Terms: interventions — palbociclib; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Two-Period Fixed-Sequence Arm (Experimental): This arm is comprised of two treatment periods in fixed sequence. Period 1 is 7 days long, while Period 2 is 28 days long. In Period 1 the subjects receive a single 125 mg oral dose of PD-0332991 on Day 1. In Period 2 the subjects receive 4 daily 60 mg oral doses of tamoxifen (Days 1-4), followed by 23 daily 20 mg oral doses of tamoxifen (Days 5-27). On Day 22 of Period 2 the subjects receive a second 125 mg oral dose of PD-0332991.
  Interventions: Drug: PD-0332991 alone; Drug: Tamoxifen 60 mg; Drug: Tamoxifen 20 mg; Drug: PD-0332991 combination

INTERVENTIONS:
Drug: PD-0332991 alone — PD-0332991 is administered alone as a single oral 125 mg dose on Day 1 of Period 1.
  Other Names: PD-0332991, palbociclib
Drug: Tamoxifen 60 mg — On Days 1-4 of Period 2, tamoxifen is administered daily as 60 mg oral doses (using three 20mg tablets).
Drug: Tamoxifen 20 mg — On Days 5-27 of Period 2, tamoxifen is administered daily as 20 mg oral doses.
Drug: PD-0332991 combination — PD-0332991 is administered in combination with tamoxifen on Day 22 of Period 2 as a single 125 mg oral dose.
  Other Names: PD-0332991, palbociclib

SUMMARY:
A single 125 mg oral dose of the investigational compound PD-0332991 will be administered alone and after steady-state dosing of tamoxifen to determine if coadministration of tamoxifen alters the plasma pharmacokinetics of PD-0332991 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male between the ages of 18 and 55 years of age inclusive
* Body mass index (BMI) between 17.5 and 30.5 kg/m2
* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* a positive urine drug screen
* a supine systolic blood pressure >140 mm Hg, or diastolic blood pressure >90 mm H.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] of PD-0332991 | 0-144 hrs post PD-0332991 dose
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PD-0332991 | 0-144 hrs post PD-0332991 dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Maximum Observed Plasma Concentration (Cmax) of PD-0332991 | 0-144 hrs post PD-0332991 dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PD-0332991 | 0-144 hrs post PD-0332991 dose
Plasma Decay Half-Life (t1/2) of PD-0332991 | 0-144 hrs post PD-0332991 dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) of PD-0332991 | 0-144 hrs post PD-0332991 dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) of PD-0332991 | 0-144 hrs post PD-0332991 dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Minimum Observed Plasma Trough Concentration (Cmin) of tamoxifen | Days 1, 5, 12, 21, 22, and 28 of Period 2
Minimum Observed Plasma Trough Concentration (Cmin) of 4-hydroxytamoxifen | Days 1, 5, 12, 21, 22, and 28 of Period 2
Minimum Observed Plasma Trough Concentration (Cmin) of N-desmethyltamoxifen | Days 1, 5, 12, 21, 22, and 28 of Period 2
Minimum Observed Plasma Trough Concentration (Cmin) of endoxifen | Days 1, 5, 12, 21, 22, and 28 of Period 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481026